CLINICAL TRIAL: NCT05289687
Title: A Phase II Study of Daratumumab-Hyaluronidase for Chemotherapy-Relapsed/Refractory Minimal Residual Disease (MRD) in T Cell Acute Lymphoblastic Leukemia (T-ALL
Brief Title: Daratumumab for Chemotherapy-Refractory Minimal Residual Disease in T Cell ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA9213
Record Dates: First submitted 2022-02-18; First posted 2022-03-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: T-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — daratumumab; Hyaluronoglucosaminidase

STUDY DESIGN:
Intervention Model Description: This is a single arm study of daratumumab-hyaluronidase in T-ALL patients in morphologic CR with persistent or relapsed MRD. MRD will be assessed centrally for eligibility and response by flow cytometry. All patients will receive daratumumab-hyaluronidase once weekly for up to 4 doses during Course 1. .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Course 1 (Experimental): Daratumumab-hyaluronidase
  Interventions: Drug: Daratumumab / Hyaluronidase Injection

INTERVENTIONS:
Drug: Daratumumab / Hyaluronidase Injection — Daratumumab-hyaluronidase 1800mg/ 30,000 units once weekly for 4 doses on Days 1, 8, 15, and 22
Drug: Daratumumab / Hyaluronidase Injection — Patients that are MRD Negative on Day 29 will receive daratumumab-hyaluronidase 1800mg/ 30,000 units once weekly for 4 doses on Days 36, 43, 50, and 57.
Drug: Daratumumab / Hyaluronidase Injection — Patients that remain MRD positive on Day 29 will receive a combination of daratumumab-hyaluronidase 1800mg/ 30,000 units once weekly for 4 doses on Days 36, 43, 50, and 57 and chemotherapy selected from the combinations listed below:
  * Cytarabine 3000 mg/m2, IV, Every 12 hours for 4 doses on Days 37 and 38
  * Methotrexate 1000 mg/m2, IV, Over 24 hours on Day 36
  OR
  * Methotrexate, Starting dose 100 mg/m2, IV, Days 36, 46, 56
  * Vincristine, 1.5 mg/m2 (2 mg cap), IV, Days 36, 46, 56
  * Pegaspargase, 2000 IU/m2 (Capped at 3750 IU), IV Days 37, 57
  * Methotrexate 15 mg, IT, Days 36, 56
Drug: Daratumumab / Hyaluronidase Injection — All patients with MRD negative response after completion of previous course are eligible for daratumumab-hyaluronidase 1800mg/ 30,000 units every 2 weeks on Days 1,15, 29, 43, 57, 71, 85, and 99 for 8 doses.

SUMMARY:
In this study, the investigators are hypothesizing that daratumumab-hyaluronidase will effectively treat T-ALL in patients who have persistent or recurrent MRD following treatment with chemotherapy.

DETAILED DESCRIPTION:
The primary hypothesis is that daratumumab-hyaluronidase will effectively eliminate chemotherapy refractory and relapsed MRD in T-ALL. The secondary hypotheses include; daratumumab-hyaluronidase will improve hematologic relapse free survival (RFS),daratumumab-hyaluronidase will improve overall survival (OS), patients that achieve complete MRD response with daratumumab will have improved survival outcomes, and daratumumab-hyaluronidase will be well tolerated in T-ALL after allogenic stem cell transplant.

The primary objective of this study is to evaluate the rate of complete MRD response by flow cytometry after 4 weekly doses of daratumumab-hyaluronidase (Day 29) among patients with MRD positive T-ALL in hematologic morphologic complete remission or complete remission with incomplete hematologic recovery. The secondary objectives include; evaluation of morphologic relapse free survival (RFS), evaluation of overall survival (OS), assessment of the the survival outcomes in patients that undergo allogeneic stem cell transplant after complete MRD response with daratumumab-hyaluronidase, assessment of adverse effects and tolerability of daratumumab-hyaluronidase in T-ALL, and assessment of flow cytometry based MRD status on Day 64 of treatment or upon count recovery for patients that receive chemotherapy in addition to daratumumab-hyaluronidase during Course 1A.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have documented T cell ALL and must be in first or later hematologic CR or CRi after a minimum of 2 blocks of intensive chemotherapy.
* Patients in hematologic CR or CRi must have persistent or recurrent MRD ≥ 10-4.
* Institution must have received central MRD status test results confirming persistent or recurrent MRD ≥ 10-4 by flow cytometry.
* Patient may have undergone a prior allogeneic stem cell transplant, but patient may not have Grafts Versus Host Disease (GVHD) that requires ongoing immunosuppressive therapy. Patient may receive prednisone if the dose is ≤ 10 mg per day.
* Patient must have an ECOG performance status 0-2.
* All patients of childbearing potential must have a blood test or urine study within 14 days prior to Step 1 registration to rule out pregnancy.
* Patients must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and continue to 3 months after the last dose of protocol treatment. Patients must also agree to abstain from donating sperm, even if they have had a successful vasectomy, or donating eggs while on study treatment and for 3 months after the last dose of protocol treatment.
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
* Patient must have adequate organ and marrow function as defined below (these labs must be obtained ≤ 7 days prior to Step 1 registration).
* Absolute neutrophil count (ANC) ≥ 750/μL
* Platelets ≥ 75,000/μL
* Total or Direct bilirubin ≤ 2 mg/dL
* AST(SGOT)/ALT(SGPT) ≤ 3.0 × institutional ULN
* Creatinine ≤ 1.5 x institutional ULN or Creatinine Clearance > 30 ml/min
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with prior CNS involvement are eligible as long as they do not have active CNS involvement at time of Step 1 registration.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

Exclusion Criteria:

-Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete Remission (CR) | Day 29
  Requires that all of the following be present.
  * Peripheral Blood Counts
  * Neutrophil count ≥ 1,000/µL.
  * Platelet count ≥ 100,000/µL.
  * Reduced hemoglobin concentration or hematocrit has no bearing on remission status.
  * Leukemic blasts must not be present in the peripheral blood.
  * Bone Marrow Aspirate and Biopsy
  * Cellularity of bone marrow biopsy must be > 20% with maturation of all cell lines.
  * ≤ 5% T lymphoblasts by flow cytometry.
  * Extramedullary leukemia, such as CNS or soft tissue involvement, must not be present.
Complete Remission (CR) | Day 64
  Requires that all of the following be present.
  * Peripheral Blood Counts
  * Neutrophil count ≥ 1,000/µL.
  * Platelet count ≥ 100,000/µL.
  * Reduced hemoglobin concentration or hematocrit has no bearing on remission status.
  * Leukemic blasts must not be present in the peripheral blood.
  * Bone Marrow Aspirate and Biopsy
  * Cellularity of bone marrow biopsy must be > 20% with maturation of all cell lines.
  * ≤ 5% T lymphoblasts by flow cytometry.
  * Extramedullary leukemia, such as CNS or soft tissue involvement, must not be present.
Complete Response with Partial Count Recovery (CRh) | Day 29
  The same as for CR except with unsupported platelets > 50,000/μL, hemoglobin > 7 g/dL, and absolute neutrophil count > 500/μL.
Complete Response with Partial Count Recovery (CRh) | Day 64
  The same as for CR except with unsupported platelets > 50,000/μL, hemoglobin > 7 g/dL, and absolute neutrophil count > 500/μL.
Complete Remission incomplete (CRi) | Day 29
  All the same response criteria in peripheral blood and bone marrow as CR with the exception that there is incomplete platelet recovery (platelets > 75,000/uL but < 100,000/μL independent of platelet transfusions) or incomplete neutrophil count recovery > 750/uL but < 1000/μL.
Complete Remission incomplete (CRi) | Day 64
  All the same response criteria in peripheral blood and bone marrow as CR with the exception that there is incomplete platelet recovery (platelets > 75,000/uL but < 100,000/μL independent of platelet transfusions) or incomplete neutrophil count recovery > 750/uL but < 1000/μL.
Minimal Residual Disease Negativity (MRD-) | Day 29
  Bone marrow lymphoblast percent < 0.01% (< 10-4) by flow cytometry in a patient that fulfills count requirements for CR/CRh/CRi..
Minimal Residual Disease Negativity (MRD-) | Day 64
  Bone marrow lymphoblast percent < 0.01% (< 10-4) by flow cytometry in a patient that fulfills count requirements for CR/CRh/CRi..
Morphologic Relapse | Day 29
  Bone Marrow Aspirate and Biopsy
  * Presence of > 5% T lympho-blasts, not attributable to another cause (e.g., bone marrow regeneration).
  * If there are no circulating blasts and the bone marrow contains 5% to 20% blasts, then a repeat bone marrow performed ≥ 1 week later documenting more than 5% blasts is necessary to meet the criteria for relapse.
MRD Relapse | Day 29
  • Relapse following MRD negativity is defined as bone marrow T lymphoblast percent ≥ 0.01% (10-4).
Morphologic Relapse | Day 64
  Bone Marrow Aspirate and Biopsy
  * Presence of > 5% T lympho-blasts, not attributable to another cause (e.g., bone marrow regeneration).
  * If there are no circulating blasts and the bone marrow contains 5% to 20% blasts, then a repeat bone marrow performed ≥ 1 week later documenting more than 5% blasts is necessary to meet the criteria for relapse.
MRD Relapse | Day 64
  • Relapse following MRD negativity is defined as bone marrow T lymphoblast percent ≥ 0.01% (10-4).
Refractory | Day 29
  Failure to achieve MRD negativity as defined by bone marrow with CR/CRh/CRi with T lymphoblast percent ≥ 0.01% (10-4).
Refractory | Day 64
  Failure to achieve MRD negativity as defined by bone marrow with CR/CRh/CRi with T lymphoblast percent ≥ 0.01% (10-4).

CONTACTS AND LOCATIONS:
Overall Officials: Shira Dinner, MD, Study Chair — Northwestern University
Locations (1):
- Northwestern, Chicago, Illinois, United States

REFERENCES:
- [Background] Dores GM, Devesa SS, Curtis RE, Linet MS, Morton LM. Acute leukemia incidence and patient survival among children and adults in the United States, 2001-2007. Blood. 2012 Jan 5;119(1):34-43. doi: 10.1182/blood-2011-04-347872. Epub 2011 Nov 15. PMID 22086414
- [Background] Hunger SP, Lu X, Devidas M, Camitta BM, Gaynon PS, Winick NJ, Reaman GH, Carroll WL. Improved survival for children and adolescents with acute lymphoblastic leukemia between 1990 and 2005: a report from the children's oncology group. J Clin Oncol. 2012 May 10;30(14):1663-9. doi: 10.1200/JCO.2011.37.8018. Epub 2012 Mar 12. PMID 22412151
- [Background] Steinherz PG, Gaynon PS, Breneman JC, Cherlow JM, Grossman NJ, Kersey JH, Johnstone HS, Sather HN, Trigg ME, Uckun FM, Bleyer WA. Treatment of patients with acute lymphoblastic leukemia with bulky extramedullary disease and T-cell phenotype or other poor prognostic features: randomized controlled trial from the Children's Cancer Group. Cancer. 1998 Feb 1;82(3):600-12. doi: 10.1002/(sici)1097-0142(19980201)82:33.0.co;2-4. PMID 9452280
- [Background] Marks DI, Paietta EM, Moorman AV, Richards SM, Buck G, DeWald G, Ferrando A, Fielding AK, Goldstone AH, Ketterling RP, Litzow MR, Luger SM, McMillan AK, Mansour MR, Rowe JM, Tallman MS, Lazarus HM. T-cell acute lymphoblastic leukemia in adults: clinical features, immunophenotype, cytogenetics, and outcome from the large randomized prospective trial (UKALL XII/ECOG 2993). Blood. 2009 Dec 10;114(25):5136-45. doi: 10.1182/blood-2009-08-231217. PMID 19828704
- [Background] Schrappe M, Valsecchi MG, Bartram CR, Schrauder A, Panzer-Grumayer R, Moricke A, Parasole R, Zimmermann M, Dworzak M, Buldini B, Reiter A, Basso G, Klingebiel T, Messina C, Ratei R, Cazzaniga G, Koehler R, Locatelli F, Schafer BW, Arico M, Welte K, van Dongen JJ, Gadner H, Biondi A, Conter V. Late MRD response determines relapse risk overall and in subsets of childhood T-cell ALL: results of the AIEOP-BFM-ALL 2000 study. Blood. 2011 Aug 25;118(8):2077-84. doi: 10.1182/blood-2011-03-338707. Epub 2011 Jun 30. PMID 21719599
- [Background] Beldjord K, Chevret S, Asnafi V, Huguet F, Boulland ML, Leguay T, Thomas X, Cayuela JM, Grardel N, Chalandon Y, Boissel N, Schaefer B, Delabesse E, Cave H, Chevallier P, Buzyn A, Fest T, Reman O, Vernant JP, Lheritier V, Bene MC, Lafage M, Macintyre E, Ifrah N, Dombret H; Group for Research on Adult Acute Lymphoblastic Leukemia (GRAALL). Oncogenetics and minimal residual disease are independent outcome predictors in adult patients with acute lymphoblastic leukemia. Blood. 2014 Jun 12;123(24):3739-49. doi: 10.1182/blood-2014-01-547695. Epub 2014 Apr 16. PMID 24740809
- [Background] Bruggemann M, Raff T, Flohr T, Gokbuget N, Nakao M, Droese J, Luschen S, Pott C, Ritgen M, Scheuring U, Horst HA, Thiel E, Hoelzer D, Bartram CR, Kneba M; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Clinical significance of minimal residual disease quantification in adult patients with standard-risk acute lymphoblastic leukemia. Blood. 2006 Feb 1;107(3):1116-23. doi: 10.1182/blood-2005-07-2708. Epub 2005 Sep 29. PMID 16195338
- [Background] Gokbuget N, Kneba M, Raff T, Trautmann H, Bartram CR, Arnold R, Fietkau R, Freund M, Ganser A, Ludwig WD, Maschmeyer G, Rieder H, Schwartz S, Serve H, Thiel E, Bruggemann M, Hoelzer D; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Adult patients with acute lymphoblastic leukemia and molecular failure display a poor prognosis and are candidates for stem cell transplantation and targeted therapies. Blood. 2012 Aug 30;120(9):1868-76. doi: 10.1182/blood-2011-09-377713. Epub 2012 Mar 22. PMID 22442346
- [Background] Teachey DT, Hunger SP. Predicting relapse risk in childhood acute lymphoblastic leukaemia. Br J Haematol. 2013 Sep;162(5):606-20. doi: 10.1111/bjh.12442. Epub 2013 Jun 29. PMID 23808872
- [Background] Brent L. Wood, Stuart S. Winter, Kimberly P. Dunsmore, Meenakshi Devidas, Si Chen, Barbara Asselin, Natia Esiashvili, Mignon L. Loh, Naomi J. Winick, William L. Carroll, Elizabeth A. Raetz SPH. T-lymphoblastic leukemia (T-ALL) shows excellent outcome, lack of significance of the early Thymic precursor (ETP) Immunophenotype, and validation of the prognostic value of end- induction minimal residual disease (MRD) in Children's oncology group (COG) Study AALL0434 Blood 2014;124.
- [Background] Wood BL, Winter SS, Dunsmore KP, Devidas M, Chen S, Asselin B, et al. Patients with early T-cell precursor (ETP) acute lymphoblastic leukemia (ALL) have high levels of minimal residual disease (MRD) at the end of induction-a Children's oncology group (COG) study [abstract]. Blood. 2009;114.
- [Background] Quist-Paulsen P, Toft N, Heyman M, Abrahamsson J, Griskevicius L, Hallbook H, Jonsson OG, Palk K, Vaitkeviciene G, Vettenranta K, Asberg A, Frandsen TL, Opdahl S, Marquart HV, Siitonen S, Osnes LT, Hultdin M, Overgaard UM, Wartiovaara-Kautto U, Schmiegelow K. T-cell acute lymphoblastic leukemia in patients 1-45 years treated with the pediatric NOPHO ALL2008 protocol. Leukemia. 2020 Feb;34(2):347-357. doi: 10.1038/s41375-019-0598-2. Epub 2019 Oct 14. PMID 31611626
- [Background] Gokbuget N, Dombret H, Bonifacio M, Reichle A, Graux C, Faul C, Diedrich H, Topp MS, Bruggemann M, Horst HA, Havelange V, Stieglmaier J, Wessels H, Haddad V, Benjamin JE, Zugmaier G, Nagorsen D, Bargou RC. Blinatumomab for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukemia. Blood. 2018 Apr 5;131(14):1522-1531. doi: 10.1182/blood-2017-08-798322. Epub 2018 Jan 22. PMID 29358182
- [Background] Bride KL, Vincent TL, Im SY, Aplenc R, Barrett DM, Carroll WL, Carson R, Dai Y, Devidas M, Dunsmore KP, Fuller T, Glisovic-Aplenc T, Horton TM, Hunger SP, Loh ML, Maude SL, Raetz EA, Winter SS, Grupp SA, Hermiston ML, Wood BL, Teachey DT. Preclinical efficacy of daratumumab in T-cell acute lymphoblastic leukemia. Blood. 2018 Mar 1;131(9):995-999. doi: 10.1182/blood-2017-07-794214. Epub 2018 Jan 5. PMID 29305553
- [Background] Vogiatzi F, Winterberg D, Lenk L, Buchmann S, Cario G, Schrappe M, Peipp M, Richter-Pechanska P, Kulozik AE, Lentes J, Bergmann AK, Valerius T, Frielitz FS, Kellner C, Schewe DM. Daratumumab eradicates minimal residual disease in a preclinical model of pediatric T-cell acute lymphoblastic leukemia. Blood. 2019 Aug 22;134(8):713-716. doi: 10.1182/blood.2019000904. Epub 2019 Jul 16. No abstract available. PMID 31311816
- [Background] Ofran Y, Ringelstein-Harlev S, Slouzkey I, Zuckerman T, Yehudai-Ofir D, Henig I, Beyar-Katz O, Hayun M, Frisch A. Daratumumab for eradication of minimal residual disease in high-risk advanced relapse of T-cell/CD19/CD22-negative acute lymphoblastic leukemia. Leukemia. 2020 Jan;34(1):293-295. doi: 10.1038/s41375-019-0548-z. Epub 2019 Aug 21. No abstract available. PMID 31435023
- [Background] Fulcher J, Berardi P, Christou G, Villeneuve PJA, Bredeson C, Sabloff M. Nelarabine-containing regimen followed by daratumumab as an effective salvage therapy and bridge to allogeneic hematopoietic stem cell transplantation for primary refractory early T-cell precursor lymphoblastic leukemia. Leuk Lymphoma. 2021 Sep;62(9):2295-2297. doi: 10.1080/10428194.2021.1901097. Epub 2021 Mar 21. No abstract available. PMID 33749497
- [Background] Ruhayel SD, Valvi S. Daratumumab in T-cell acute lymphoblastic leukaemia: A case report and review of the literature. Pediatr Blood Cancer. 2021 May;68(5):e28829. doi: 10.1002/pbc.28829. Epub 2020 Nov 27. No abstract available. PMID 33245179
- [Background] Cerrano M, Castella B, Lia G, Olivi M, Faraci DG, Butera S, Martella F, Scaldaferri M, Cattel F, Boccadoro M, Massaia M, Ferrero D, Bruno B, Giaccone L. Immunomodulatory and clinical effects of daratumumab in T-cell acute lymphoblastic leukaemia. Br J Haematol. 2020 Oct;191(1):e28-e32. doi: 10.1111/bjh.16960. Epub 2020 Jul 19. No abstract available. PMID 32686081
- [Background] Mirgh S, Ahmed R, Agrawal N, Khushoo V, Garg A, Francis S, Tejwani N, Singh N, Bhurani D. Will Daratumumab be the next game changer in early thymic precursor-acute lymphoblastic leukaemia? Br J Haematol. 2019 Oct;187(2):e33-e35. doi: 10.1111/bjh.16154. Epub 2019 Aug 26. No abstract available. PMID 31452197
- [Background] Bonda A, Punatar S, Gokarn A, Mohite A, Shanmugam K, Nayak L, Bopanna M, Cheriyalinkal Parambil B, Khattry N. Daratumumab at the frontiers of post-transplant refractory T-acute lymphoblastic leukemia-a worthwhile strategy? Bone Marrow Transplant. 2018 Nov;53(11):1487-1489. doi: 10.1038/s41409-018-0222-5. Epub 2018 Jun 8. No abstract available. PMID 29884853
- [Background] Mateos MV, Nahi H, Legiec W, Grosicki S, Vorobyev V, Spicka I, Hungria V, Korenkova S, Bahlis N, Flogegard M, Blade J, Moreau P, Kaiser M, Iida S, Laubach J, Magen H, Cavo M, Hulin C, White D, De Stefano V, Clemens PL, Masterson T, Lantz K, O'Rourke L, Heuck C, Qin X, Parasrampuria DA, Yuan Z, Xu S, Qi M, Usmani SZ. Subcutaneous versus intravenous daratumumab in patients with relapsed or refractory multiple myeloma (COLUMBA): a multicentre, open-label, non-inferiority, randomised, phase 3 trial. Lancet Haematol. 2020 May;7(5):e370-e380. doi: 10.1016/S2352-3026(20)30070-3. Epub 2020 Mar 23. PMID 32213342
- [Background] Short N, Kantarjian H, Patel K, et al. Ultrasensitive Next-Generation Sequencing-Based Measurable Residual Disease Assessment in Philadelphia Chromosome-Negative Acute Lymphoblastic Leukemia after Frontline Therapy: Correlation with Flow Cytometry and Impact on Clinical Outcomes. Blood. 2020 Nov 5; 136(1): Abstract 583.
- [Background] Muffly L, Sundaram V, Chen C, et al. Monitoring Measurable Residual Disease Using Peripheral Blood in Acute Lymphoblastic Leukemia: Results of a Prospective, Observational Study. Blood. 2020 Nov 5; 136(1): Abstract 975.